CLINICAL TRIAL: NCT04217603
Title: Effect of Continuous Positive Airway Pressure (CPAP) on 6-Minute Walk Test Outcomes in Patients With Excessive Central Airway Collapse (ECAC)
Brief Title: Effect of CPAP on 6-Minute Walk Test Outcomes in Patients With ECAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief, Section of Interventional Pulmonology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P001034
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Tracheobronchomalacia; Excessive Dynamic Airway Collapse
Keywords: Continuous Positive Airway Pressure; Tracheobronchomalacia; Excessive Dynamic Airway Collapse; Excessive Central Airway Collapse
MeSH Terms: conditions — Tracheobronchomalacia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: This prospective, randomized placebo controlled, double-blind clinical trial will be conducted at Beth Israel Deaconess Medical Center (BIDMC) in accordance with Good Clinical Practice Standards and under IRB supervision. We plan to enroll a total of 32 patients with ECAC randomized by an opaque envelope technique into two different groups: group 1 (CPAP) and group 2 (sham-CPAP)
  * Group 1: This group will perform a 6MWT with CPAP
  * Group 2: This group will perform a 6MWT with a sham-CPAP
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be stratified using the variables sex (Female and male) and age (<60 and >60). Additionally a block 2-4 pattern will be used to assure a random and evenly distributed patient population in the different strata. Randomization will be carried out by the research coordinator; the rest of the personnel will be blinded to the allocation of the patients to the different groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): This group will perform a 6MWT with CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP) device
- Group 2 (Sham Comparator): This group will perform a 6MWT with a sham-CPAP
  Interventions: Device: Sham-continuous positive airway pressure (CPAP) device

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) device — Use of a CPAP during a 6 minute walk test to maintain the airways open during the respiratory cycle
  Arms: Group 1
Device: Sham-continuous positive airway pressure (CPAP) device — An enlarged air leak incorporated into the exhalation valve will be positioned between the mask and the CPAP tubing, allowing airflow resistance of the exhalation port to be almost eliminated by increasing its area, thereby virtually cancelling positive pressure. Also an orifice restrictor in the CPAP circuit will be connected between the CPAP unit and the tubing in order to load the blower with the same airflow resistance as in true CPAP.
  Arms: Group 2

SUMMARY:
The purpose of this protocol is to perform a prospective, randomized, double-blinded, pacebo-controlled clinical trial to determine the influence of a non-invasive positive pressure ventilation device on exercise capacity and symptoms in adult patients with ECAC. Primary outcome will include the total distance traversed by the study subject during a standard 6-minute walk test, and secondary outcomes will include peak flow measurement and symptom reporting before and after the exercise testing. The study will focus on the use of continuous positive airway pressure (CPAP) device. CPAP is FDA-approved for the treatment of various medical conditions, including obstructive sleep apnea and heart failure, but is not FDA-approved for the treatment of ECAC. The study will enroll 32 ambulatory study subjects with confirmed ECAC at the BIDMC, and each study subject will be monitored for up to 3 months.

DETAILED DESCRIPTION:
Basal 6MWT performed as a standard of care in these patients will be compared to intervention ones to see if there is an improvement of at least 24 meters in their 6MWT distance, then both groups will be compared to see if there is a statistically significant difference between groups. Subjects, treating physicians and the research fellow performing the 6MWT will be blinded to the intervention; the only un-blinded personnel to the intervention will be the study coordinator who will be in charge of setting the CPAP before every intervention.

As part of the standard of care of our institution, patients that are referred due to suspicion of ECAC undergo initial PFTs, 6MWT and dynamic CT scan. With this information, patients are evaluated in clinic by the interventional pulmonary and thoracic surgery team who decide if the patient has the mentioned disease based on the previous testing. To corroborate the findings patients with moderate so severe disease are taken into a bronchoscopy with dynamic maneuvers as part of the standard of care. Initial bronchoscopic examination will be performed as described in the following section "I-Dynamic Bronchoscopy Protocol" as part of the standard of care of patients. After initial evaluation, during the same intervention, all patients that agree to participate in our study will go through a CPAP calibration procedure; in order to determine the adequate pressure to achieve airway patency of at least 70% during end exhalation in each individual case. After regular bronchoscopic examination, a full face F&P SimplusTM CPAP mask (Fisher & Paykel, Irvine, CA, USA) will be placed in all patients to prevent un-blinding the treating physician. The mask will be connected to a dual axis swivel adapter (T-adapter) and the bronchoscope will be advanced to the nares through the swivel adaptor; air leak will be prevented by the tight disposable cap of the swivel adaptor as described by Murgu et al.20

The calibration process will be performed following the technique first described by Ferguson et al10, bronchoscope will be positioned to assess the area with ECAC previously identified during regular examination; bronchoscope will be placed in the center of the lumen while assuring a constant 1-cm distance between the tip of the bronchoscope and the target area being measured, images will be taken during end inspiration and end expiration, gradual increases of 1 cmH2O in the CPAP pressure will be made until a 70% or less collapse is seen during end expiration by the bronchoscopist. At any given pressure increase the assessment of airway collapse will be made in 3 different respiratory cycles, the whole procedure will be recorded and posteriorly analyzed using morphometric bronchoscopy (Image J analysis program) as described in the "Morphometric Bronchoscopy" section.

Patient Population Subjects (>18 years of age) with previous diagnosis of ECAC confirmed by dynamic CT scan and/or bronchoscopy, who are currently receiving adequate medical therapy (Optimal medication doses and interventions defined by Interventional Pulmonary team) for comorbidities such as COPD, GERD, asthma, etc and are able to perform a 6 MWT.

Tracheobronchomalacia Evaluation CT Central Airway Protocol: All patients will be imaged according to our standard low dose CT central airway protocol21, which includes imaging during end-inspiratory and continuous dynamic expiratory phases. A multidetector row, helical CT scanner (LightSpeed; GE Medical Systems; Milwaukee, WI; or Aquilion; Toshiba America Medical Systems; Tustin, CA) which includes 4, 8, 16, and 64 detector-row systems will be used. Helical scanning will be performed in the cranio-caudal dimension during both respiratory phases. An experienced thoracic radiologist will review the CT images on a picture archiving and communication system (PACS) [Path-Speed, General Electric Medical Systems]. Using a computerized tracing tool in our PACS system, the inner wall of the airway will be hand traced at the level of maximal collapse in dynamic expiratory images to calculate the cross-sectional area of the airway (mm2). At the same level on end-inspiration images, the cross-sectional area of the airway lumen will be determined by using the same method. The percentage of luminal collapse between both respiratory phases will be calculated using the following formula= [1 - (Aee/Aei)],) X100, where Aee is luminal area at end expiration and Aei is luminal area at end inspiration. Mild ECAC is diagnosed if the percent of luminal collapse during dynamic expiration is 70-80%, moderate from 80-90% and severe >90%.

I-Dynamic Bronchoscopy Protocol All patients who are enrolled for the study will undergo bronchoscopy under minimal sedation using intravenous midazolam and fentanyl to allow spontaneous respiration. Lidocaine (1%, 20 ml), will be delivered by atomizer to the posterior oropharynx until the gag reflex is suppressed. The larynx, vocal cords, aryepiglottic folds and entire tracheobronchial tree will be irrigated with 1% lidocaine in 2-ml aliquots delivered through the bronchoscope during the procedure. An Olympus BF P180 video bronchoscope (Olympus America, Melville, NY) with a 4.9-mm outer diameter and 2.0-mm working channel will be used to minimize any stenting effect. The bronchoscope will be introduced into the proximal trachea at the level of the cricoid. At that point, patients will be instructed to take a deep breath, hold it and then blow it out (forced expiratory maneuver). Maneuver will be done at the following six sites: proximal trachea at the level of the cricoid; mid-trachea 5 cm proximal to the carina; distal trachea 2 cm proximal to the carina; right main stem bronchus at the right tracheobronchial angle; bronchus intermedius and left main bronchus at the left tracheobronchial angle. The maneuver will be repeated three times to ensure maximal airway narrowing during exhalation. All bronchoscopies will be video recorded and reviewed after the procedure to assess the degree of airway collapse. Mild ECAC is defined as a collapse 70-80%, moderate 80-90% and severe >90% of the airway during exhalation. This is standard of care for patients with EDAC.

After collapse degree is assessed trough forced expiratory maneuver, a nasal CPAP device (Define model) will be used in the patient, forced expiratory maneuvers will be repeated with different CPAP configurations until a 70% or less airway collapse is achieved. Calibration at which 70% airway collapse is achieved will be recorded and posteriorly used as the CPAP volume for the second 6MWT.

Morphometric bronchoscopy Cross-sectional area (CSA) of the airway will be calculated after the procedure by using the Image J analysis program (available free of charge at http://rsb.info.nih.gov/ij/) using two different measurement techniques as it was described by Murgu et al.22 The graphical measurement method uses color levels within the image to identify an appropriate region to be measured. Images are imported into Image J and a color balance window is opened (Image > Adjust > Color Balance). The histogram is then set to RGB color. The minimum and maximum bars are adjusted so that the resulting line corresponds to the highest point of the histogram. Only red, yellow, white, and black colors then remain. The black area, which represents the region to be measured for CSA, is selected using a wand tool. Using the region of interest (ROI) Manager (Analyze > Tools > ROI Manager) the selected area is then calculated in pixels. The manual measurement method requires that the operator selects the area to be measured by first opening the image using Image J. Using the polygon selections tool, the area of interest is then selected, and the ROI manager is used as in the graphical method.

Finally to provide an objective measurement in our patients, a collapsibility index (CI) will be calculated: difference in airway lumen size between end inspiration and end expiration: CI = (CSAinspir - CSAexpir)/(CSAinspire x 100%). Then measurements obtained for each patient during 3 respiratory cycles will be compared to discard that there is any significant statistical difference between them.

Six Minute Walk Test The 6MWT is a test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. Testing will be performed by the study personnel in a controlled environment. Supplies such as oxygen, sublingual nitroglycerine, aspirin, and albuterol (metered dose inhaler or nebulizer) will be available. The distance walked will be reported in meters. Data from both groups will be compared in order to verify if CPAP has a positive impact on exercise capacity in these patients. Since subjects have never used CPAP before and are not used to the device a 10 minute Run-in period will be allowed in which the CPAP will be placed while the patient is seating to allow he/she to get used to the sensation generated by the machine, at this time the study personnel will also look for air leaks that could compromise the results of the study. Either a regular CPAP or a sham-CPAP will be used for the Run-in period depending on the result of the randomization; this will be done to avoid the patient noticing the difference between this period and the 6 MWT which could happen if only regular CPAP was used.

Sham-CPAP The Sham-CPAP will be created following the methods of Farre et al23 And Rodway et al.24 An enlarged air leak incorporated into the exhalation valve will be positioned between the mask and the CPAP tubing, allowing airflow resistance of the exhalation port to be almost eliminated by increasing its area, thereby virtually cancelling positive pressure. Also an orifice restrictor in the CPAP circuit will be connected between the CPAP unit and the tubing in order to load the blower with the same airflow resistance as in true CPAP. These changes allow the ventilator operating noise and the airflow through the exhalation port remain unchanged, which are crucial to a CPAP placebo.

Enrollment CPAP naïve patients with a diagnosis of ECAC will be informed about the trial and if interested will be recruited for our randomized controlled study. Patients who meet the inclusion criteria by the principle investigator or co-investigators will be approached during an office visit to our Chest Disease Clinic at BIDMC

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of ECAC either via bronchoscopy or CT Scan
* Age > 18 years
* Patients that will undergo a diagnostic or therapeutic bronchoscopy as part of their standard of care
* Patients with a baseline 6 MWT
* Patients that have never used CPAP devices in the past

Exclusion Criteria:

* Patients with poorly-controlled respiratory comorbidities (asthma, COPD, obstructed sleep apnea, GERD, relapsing polychondritis)
* No evidence for acute respiratory tract infection, or respiratory tract infection within the prior 3 weeks
* Resting bradycardia (<50 beats/min), frequent multifocal PVCs, complex ventricular arrhythmia, sustained SVT
* Dysrhythmia that might pose a risk during exercise or training
* Any disease or condition that interferes with completion of initial or follow-up assessments
* Subject has co-morbidities that may significantly reduce subject's ability to improve exercise capacity (e.g., severe arthritis, planned knee surgery) or baseline limitation on 6MWT is not due to dyspnea.
* Subject has an inability to walk >140m (150 yd) in 6 minutes
* Subject has an inability to tolerate bronchoscopy under moderate sedation or general anesthesia.
* Subject has a known sensitivity to drugs required to perform bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Difference in meters walked in 6MWTs | 3 months
  Statistical difference between the 6 MWT results of the CPAP and sham-CPAP groups as compared with the initial results of the 6 MWT and between groups using ANCOVA.

SECONDARY OUTCOMES:
Modified Borg scale scores for dyspnea | 3 months
Modified Borg scale scores for exertion | 3 months
Subjective assestment of cough during 6MWTs | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leong P, Bardin PG, Lau KK. What's in a name? Expiratory tracheal narrowing in adults explained. Clin Radiol. 2013 Dec;68(12):1268-75. doi: 10.1016/j.crad.2013.06.017. Epub 2013 Aug 13. PMID 23953005
- [Background] Murgu S, Colt H. Tracheobronchomalacia and excessive dynamic airway collapse. Clin Chest Med. 2013 Sep;34(3):527-55. doi: 10.1016/j.ccm.2013.05.003. Epub 2013 Jun 27. PMID 23993822
- [Background] Ridge CA, O'donnell CR, Lee EY, Majid A, Boiselle PM. Tracheobronchomalacia: current concepts and controversies. J Thorac Imaging. 2011 Nov;26(4):278-89. doi: 10.1097/RTI.0b013e3182203342. PMID 22009081
- [Background] Park JG, Edell ES. Dynamic Airway Collapse: Distinct From Tracheomalacia. J Bronchol. 2005;12(3):143-146. doi:10.1097/01.laboratory.0000171764.65217.f8
- [Background] Boiselle PM, O'Donnell CR, Bankier AA, Ernst A, Millet ME, Potemkin A, Loring SH. Tracheal collapsibility in healthy volunteers during forced expiration: assessment with multidetector CT. Radiology. 2009 Jul;252(1):255-62. doi: 10.1148/radiol.2521081958. Epub 2009 May 6. PMID 19420322
- [Background] Majid A, Fernandez L, Fernandez-Bussy S, Herth F, Ernst A. [Tracheobronchomalacia]. Arch Bronconeumol. 2010 Apr;46(4):196-202. doi: 10.1016/j.arbres.2009.10.011. Epub 2009 Dec 9. Spanish. PMID 20004507
- [Background] Cepeda S, Climent M, Martinez Moragon E. [Bronchomalacia in adults: an infrequent entity that improves with continuous positive pressure on the airway]. An Sist Sanit Navar. 2016 Dec 30;39(3):457-458. doi: 10.23938/ASSN.0230. No abstract available. Spanish. PMID 28032884
- [Background] Sala A, Martínez Deltoro A, Martínez Moragón E. Asmática con broncomalacia y buena respuesta al tratamiento con presión positiva continua en la vía aérea. Arch Bronconeumol. http://www.archbronconeumol.org/es/pdf/S030028961300272X/S300/.
- [Background] Adliff M, Ngato D, Keshavjee S, Brenaman S, Granton JT. Treatment of diffuse tracheomalacia secondary to relapsing polychondritis with continuous positive airway pressure. Chest. 1997 Dec;112(6):1701-4. doi: 10.1378/chest.112.6.1701. PMID 9404780
- [Background] Ferguson GT, Benoist J. Nasal continuous positive airway pressure in the treatment of tracheobronchomalacia. Am Rev Respir Dis. 1993 Feb;147(2):457-61. doi: 10.1164/ajrccm/147.2.457. PMID 8430971
- [Background] Jiang AG, Gao XY, Lu HY. Diagnosis and management of an elderly patient with severe tracheomalacia: A case report and review of the literature. Exp Ther Med. 2013 Sep;6(3):765-768. doi: 10.3892/etm.2013.1195. Epub 2013 Jul 2. PMID 24137262
- [Background] Kandaswamy C, Balasubramanian V. Review of adult tracheomalacia and its relationship with chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2009 Mar;15(2):113-9. doi: 10.1097/MCP.0b013e328321832d. PMID 19532025
- [Background] Carden KA, Boiselle PM, Waltz DA, Ernst A. Tracheomalacia and tracheobronchomalacia in children and adults: an in-depth review. Chest. 2005 Mar;127(3):984-1005. doi: 10.1378/chest.127.3.984. PMID 15764786
- [Background] Murgu SD, Colt HG. Treatment of adult tracheobronchomalacia and excessive dynamic airway collapse : an update. Treat Respir Med. 2006;5(2):103-15. doi: 10.2165/00151829-200605020-00004. PMID 16512691
- [Background] Murgu SD. Pneumatic stenting for tracheobronchomalacia. J Bronchology Interv Pulmonol. 2014 Apr;21(2):109-12. doi: 10.1097/LBR.0000000000000053. No abstract available. PMID 24739682
- [Background] Martin JG, Shore S, Engel LA. Effect of continuous positive airway pressure on respiratory mechanics and pattern of breathing in induced asthma. Am Rev Respir Dis. 1982 Nov;126(5):812-7. doi: 10.1164/arrd.1982.126.5.812. PMID 6216839
- [Background] Smith TC, Marini JJ. Impact of PEEP on lung mechanics and work of breathing in severe airflow obstruction. J Appl Physiol (1985). 1988 Oct;65(4):1488-99. doi: 10.1152/jappl.1988.65.4.1488. PMID 3053583
- [Background] Kaltsakas G, Patout M, Arbane G, et al. Review of adult tracheomalacia and its relationship with chronic obstructive pulmonary disease. December 2017:A80-A81. doi:10.1136/thoraxjnl-2017-210983.140
- [Background] Patout M, Mylott L, Kent R, Arbane G, Murphy PB, Hart N. Trial of Portable Continuous Positive Airway Pressure for the Management of Tracheobronchomalacia. Am J Respir Crit Care Med. 2016 May 15;193(10):e57. doi: 10.1164/rccm.201511-2243IM. No abstract available. PMID 26982389
- [Background] Murgu SD, Pecson J, Colt HG. Bronchoscopy during noninvasive ventilation: indications and technique. Respir Care. 2010 May;55(5):595-600. PMID 20420731
- [Background] Zhang J, Hasegawa I, Feller-Kopman D, Boiselle PM. 2003 AUR Memorial Award. Dynamic expiratory volumetric CT imaging of the central airways: comparison of standard-dose and low-dose techniques. Acad Radiol. 2003 Jul;10(7):719-24. doi: 10.1016/s1076-6332(03)80117-4. PMID 12862281
- [Background] Murgu S, Colt HG. Morphometric bronchoscopy in adults with central airway obstruction: case illustrations and review of the literature. Laryngoscope. 2009 Jul;119(7):1318-24. doi: 10.1002/lary.20478. PMID 19444886
- [Background] Farre R, Hernandez L, Montserrat JM, Rotger M, Ballester E, Navajas D. Sham continuous positive airway pressure for placebo-controlled studies in sleep apnoea. Lancet. 1999 Apr 3;353(9159):1154. doi: 10.1016/S0140-6736(99)01056-9. No abstract available. PMID 10209985
- [Background] Rodway GW, Weaver TE, Mancini C, Cater J, Maislin G, Staley B, Ferguson KA, George CF, Schulman DA, Greenberg H, Rapoport DM, Walsleben JA, Lee-Chiong T, Kuna ST. Evaluation of sham-CPAP as a placebo in CPAP intervention studies. Sleep. 2010 Feb;33(2):260-6. doi: 10.1093/sleep/33.2.260. PMID 20175410
- [Background] Puhan MA, Chandra D, Mosenifar Z, Ries A, Make B, Hansel NN, Wise RA, Sciurba F; National Emphysema Treatment Trial (NETT) Research Group. The minimal important difference of exercise tests in severe COPD. Eur Respir J. 2011 Apr;37(4):784-90. doi: 10.1183/09031936.00063810. Epub 2010 Aug 6. PMID 20693247